CLINICAL TRIAL: NCT03897751
Title: A Safety and Effectiveness Study of a New Contact Lens Cleaning and Disinfecting Solution
Brief Title: A Safety and Effectiveness Study of BL-ABT12 Multi-Purpose Solution for Use by Participants With Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 932
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Contact Lens Wear
Keywords: Contact Lens Cleaning Solution; Disinfectants, Contact Lens; Soft Contact Lens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ABT12 Multi-Purpose Solution (Experimental): Participants will use ABT12 Multi-Purpose Solution to clean their contact lenses daily for 3 months. Participants will use Sensitive Eyes Rewetting Drops as needed during the study.
  Interventions: Device: ABT12 Multi-Purpose Solution; Device: Sensitive Eyes® Rewetting Drops
- COMPLETE Multi-Purpose Solution (Active Comparator): Participants will use COMPLETE Multi-Purpose Solution to clean their contact lenses daily for 3 months. Participants will use Sensitive Eyes Rewetting Drops as needed during the study.
  Interventions: Device: COMPLETE Multi-Purpose Solution; Device: Sensitive Eyes® Rewetting Drops

INTERVENTIONS:
Device: ABT12 Multi-Purpose Solution — Contact lens cleaning and disinfecting solution
  Arms: ABT12 Multi-Purpose Solution
Device: COMPLETE Multi-Purpose Solution — Contact lens cleaning and disinfecting solution
  Other Names: COMPLETE® Multi-Purpose Solution Easy Rub® Formula
  Arms: COMPLETE Multi-Purpose Solution
Device: Sensitive Eyes® Rewetting Drops — For use as needed during the study.

SUMMARY:
This study is to evaluate the safety and effectiveness of ABT12 Multi-Purpose solution (Test) compared to COMPLETE® Multi-Purpose Solution Easy Rub® Formula ("COMPLETE Multi-Purpose Solution") when used by participants who are habitual contact lens wearers.

DETAILED DESCRIPTION:
Eligible participants will be enrolled from 1 of 5 lens groups based on their habitual contact lenses. Participants will be randomized on a 1:1 basis within each group per site to receive either ABT12 Multi-Purpose solution or COMPLETE Multi-Purpose Solution. The 5 lens groups will be comprised of habitual wearers of soft lenses based on the following lens material:

* Etaficon A, Acuvue2, Vistakon
* Balafilcon A, PureVision2, Bausch + Lomb
* Samfilcon A, Ultra, Bausch + Lomb
* Lotrafilcon B, Optix Aqua, Alcon
* Senofilcon C, Vita, Vistakon

ELIGIBILITY:
Inclusion Criteria:

* Is able to read, understand, and provide written informed consent on the Institutional Review Board (IRB) approved Informed Consent Form (ICF) and provide authorization as appropriate local privacy regulations
* Is a habitual wearer (at least 3 months) of one of the following lens types: 1) Etaficon A, Acuvue2, Vistakon; 2) Balafilcon A, PureVision2, Bausch + Lomb; 3) Samfilcon A, Ultra, Bausch + Lomb; 4) Lotrafilcon B, Optix Aqua, Alcon; 5) Senofilcon C, Vita, Vistakon
* Vision is correctable through spherocylindrical refraction to 32 letters (0.3 logarithm of the minimum angle of resolution [logMAR]) or better (distance, high contrast) in each eye with soft spherical contact lenses
* Has clear central corneas and is free of any anterior segment disorders
* Is a habitual user of a lens care product for cleaning, disinfecting, and storage of lenses
* Requires lens correction in both eyes
* Wears the same manufacturer and brand of lens in both eyes
* Agrees to wear study lenses on a daily wear basis for approximately 3 months
* Is willing and able to comply with all treatment and follow-up/study procedures

Exclusion Criteria:

* Participants who currently use a hydrogen-peroxide cleaning and disinfecting solution
* Participating in any drug or device clinical investigation within 30 days prior to entry into this study and/or during the period of study participation
* Females of childbearing potential (those who are not surgically sterilized or postmenopausal), if they are currently pregnant, plan to become pregnant during the study, or are breastfeeding
* Has worn gas permeable (GP) lenses within the last 30 days.
* Has worn polymethylmethacrylate (PMMA) lenses within the last 3 months
* Has any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study
* Has any ocular disease or is using any ocular medication
* Is using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance
* Currently wears monovision, multifocal, or toric contact lenses
* Has ocular astigmatism of 1.00 diopter (D) or greater in either eye
* Vision is not correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye with soft spherical contact lenses
* Has anisometropia (spherical equivalent) of greater than 2.00D
* Has any Grade 2 or greater finding during the slit lamp examination
* Has corneal infiltrates, of any grade
* Participants with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear
* Has any scar or neovascularization within the central 6 millimeters (mm) of the cornea. Note that participants with minor peripheral corneal scarring (that does not extend into the central area), that, in the Investigator's judgment, does not interfere with contact lens wear, are eligible for this study
* Is aphakic
* Is amblyopic
* Has had any corneal surgery (for example, refractive surgery)
* Is allergic to any component in the study care products
* Is an employee of any of the study investigative sites or a family member of an employee of the investigative site, including family members living outside of the employee's household
* Is an Ophthalmologist, an Optometrist, an Optician, or an Ophthalmic Assistant/Technician, or currently resides with a person with any of these specialties
* Is an employee of a manufacturer of contact lenses or contact lens care products (for example, Alcon, Bausch + Lomb, Ciba Vision, CooperVision, Vistakon, or Johnson & Johnson) or currently resides with a person employed by any of these manufacturers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Bausch & Lomb Incorporated
Locations (17):
- United States (17):
  - Bausch Site 1, Birmingham, Alabama
  - Bausch Site 2, San Diego, California
  - Bausch Site 3, San Francisco, California
  - Bausch Site 4, Denver, Colorado
  - Bausch Site 5, Sarasota, Florida
  - Bausch Site 6, Decatur, Georgia
  - Bausch Site 7, Bloomington, Illinois
  - Bausch Site 9, Leavenworth, Kansas
  - Bausch Site 8, Pittsburg, Kansas
  - Bausch Site 10, Portland, Maine
  - Bausch Site 11, East Lansing, Michigan
  - Bausch Site 12, St Louis, Missouri
  - Bausch Site 13, Jamestown, New York
  - Bausch Site 14, Vestal, New York
  - Bausch Site 15, State College, Pennsylvania
  - Bausch Site 17, Brentwood, Tennessee
  - Bausch Site 16, Nashville, Tennessee

REFERENCES:
- [Derived] Schaeffer M, Shahidi A, Mosehauer G, Rah M, Reindel W. Clinical Evaluation of Biotrue Hydration Plus Multipurpose Solution in Daily Use with Planned Replacement Soft Contact Lenses. Ophthalmol Ther. 2025 Jun;14(6):1249-1260. doi: 10.1007/s40123-025-01123-0. Epub 2025 Apr 11. PMID 40216672

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT12 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution
Started | 127 | 125
Completed | 121 | 119
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT12 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution | Total
Number analyzed (Participants) | 127 | 125 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (9.72) | 34.1 (9.79) | 34.3 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 91 | 179
  Male | 39 | 34 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 10 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 101 | 103 | 204
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Overall comfort will be assessed for each eye on a scale from 0 to 100, with 100 denoting the most favorable response.
Time Frame: Month 3
Population: Randomized participants who attended the 3-month visit and did not have major protocol deviations
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | ABT12 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution
Number analyzed (Participants) | 117 | 113
Number analyzed (Eyes) | 234 | 226
score on a scale | 88.9 (11.49) | 87.5 (12.24)

2. Primary Outcome: Eye Dryness
Description: Dryness will be assessed for each eye on a scale from 0 to 100, with 100 denoting the most favorable response.
Time Frame: Month 3
Population: Randomized participants who attended the 3-month visit and did not have major protocol deviations
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | ABT12 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution
Number analyzed (Participants) | 117 | 113
Number analyzed (Eyes) | 234 | 226
score on a scale | 84.2 (15.15) | 83.1 (14.99)

3. Primary Outcome: Degree Of Lens Deposits
Description: Degree of lens deposits will be assessed for each eye as none, light, medium, or heavy.
Time Frame: Month 3
Population: Randomized participants who attended the 3-month visit and did not have major protocol deviations
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | ABT12 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution
Number analyzed (Participants) | 117 | 113
Number analyzed (Eyes) | 234 | 226
Eyes
  None or Light | 231 | 222
  Medium or Heavy | 3 | 4

4. Primary Outcome: Proportion Of Participants With Eyes With Grade >2 Slit Lamp Findings
Description: Graded slit lamp findings will be assessed for each eye using Grades 0 through 4. Greater than Grade 2 findings (Absent, Present) will be summarized at the eye level by treatment.
  Grades are 0(none), 1 (Trace), 2 (Mild), 3 (moderate), 4 (severe)
Time Frame: Day 0 (post-dispensing) through Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | ABT12 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution
Number analyzed (Participants) | 127 | 125
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | ABT12 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/125
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/125
Other Adverse Events (participants affected / at risk) | 0/127 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT03897751/Prot_SAP_000.pdf